CLINICAL TRIAL: NCT01450527
Title: Etiology and Outcomes of Acute Respiratory Distress Syndrome in Medical ICU in AIIMS
Brief Title: Etiology and Outcomes of Tropical Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, HOD Medicine, All India Institute of Medical Sciences
Other Study IDs: SKS/Med/ARDS
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Etiology and outcomes of ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient fulfilling the criteria of ARDS

SUMMARY:
This is a prospective observational study done to know the etiology and outcomes of Acute Respiratory Distress Syndrome.

DETAILED DESCRIPTION:
The study will be a prospective observational study and 64 patients with ARDS will be recruited . Written informed consent will be taken prior to inclusion of study. Study will be conducted in Medical ICU (C2 ICU) of AIIMS. Based on medical history and physical examination, radiology, biochemical and microbiological investigations etiology of ARDS will be decided.Sample will be taken at te eime of admission for estimation of inflammatory markers hsCRP,IL-1.IL-6,TNF ,Procalcitonin.From the available variables APACHE II, Sequential organ failure assessment score (SOFA), Simplified acute physiological score (SAPS)II and 3 will be calculated to assess the severity of ARDS.All patients will be given mechanical ventilation using the protocol followed by the ARDS Network low-tidal volume ventilation strategy.The data will be registered on ICU admission and there after every 24 hr. Day 0 will be defined as the interval from the time of ICU admission to 8:00 am the next day .Every day data will be recorded at a fixed time at 9 am. It will include Tidal volume Vt (ml/kg),respiratory rate/min, Minute ventilation(l/min),FiO2,PaO2/FiO2,Inspiratory flow(I:E), Ppeak (cm of H2O),Static respiratory compliance(ml/cm of water).Plateau pressure (Pplat), Peak end expiratory pressure (PEEP).Patient will be monitored throughout the course of illness and the outcome of ARDS will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fulfilling the criteria of ARDS according to American-European consensus definition
2. Admitted in medical ICU(CII/CU)
3. No known previous lung pathology e.g. bronchiectasis, Interstitial lung disease

Exclusion Criteria:

1. HIV positive serology.
2. Chronic obstructive airway disease
3. Not giving consent for study
4. Known lung pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient admitted in medical ICU
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
28-day mortality | with in 28 days after ICU admission
  Outcome(mortality) 28 days after admission

SECONDARY OUTCOMES:
Duration of hospital stay | with in the discharge from the hopsital
  Duration for which patient stays in hospital
Duration of ICU stay | Duration for which patient stays in ICU after ICU admission
  Duration for which patient stays in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K. Sharma, MD,Ph.D, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi, India